CLINICAL TRIAL: NCT00677833
Title: Phase 2/3, Open-Label, Comparative Trial Of Azithromycin Plus Chloroquine Versus Artemether-Lumefantrine For The Treatment Of Uncomplicated Plasmodium Falciparum Malaria In Children In Africa
Brief Title: Azithromycin Plus Chloroquine Versus Artemether-Lumefantrine For The Treatment Of Uncomplicated P. Falciparum Malaria In Children In Africa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0661157
Record Dates: First submitted 2008-05-12; First posted 2008-05-15 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-05

CONDITIONS: Malaria, Falciparum
Keywords: P. Falciparum Malaria; drug treatment; clinical trial
MeSH Terms: conditions — Malaria, Falciparum | interventions — Azithromycin; Chloroquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Azithromycin plus Chloroquine
- 2 (Experimental)
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Azithromycin plus Chloroquine — Combination of Azithromycin plus Chloroquine Azithromycin (~30 mg/kg) + chloroquine (~10mg base /kg) combination tablet(s) on weight basis, once daily for 3 days (Days 0,1,2) or Artemether-lumefantrine tablet(s) based on weight and labeling for 3 days (Days 0, 1, 2)
  Arms: 1
Drug: Artemether-lumefantrine — Artemether-lumefantrine tablet(s) based on weight and labeling for 3 days (Days 0, 1, 2)
  Arms: 2

SUMMARY:
The primary objective is to confirm the hypothesis that azithromycin used in combination with chloroquine is non-inferior to artemether- Lumefantrine for the treatment of symptomatic, uncomplicated malaria due to P. falciparum in children in African countries.

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys ≥5 years to ≤12 years (Cohort 1); and ≥6 to ≤59 months of age (Cohort 2) with uncomplicated, symptomatic malaria as indicated by the presence of the following:
* Blood smears positive for monoinfection with P. falciparum and asexual parasitemia between 1000 -100,000 parasites/µL;
* Documented fever (38.0°C/100.4°F rectal or tympanic; 37.2°C/99.0°F axillary or 37.5°C/99.5°F oral) or history of fever (as reported by the legally acceptable representative) within the prior 24 hours;
* Appropriate for outpatient treatment;
* Blood glucose ≥60 mg/dL;
* Hemoglobin ≥6 g/dl or hematocrit ≥18% without signs of anemia-induced Congestive Heart Failure (CHF);
* Negative urine pregnancy test for females ≥10 years of age (and of child bearing potential)

Exclusion Criteria:

* Peripheral blood smear positive for mixed infection with multiple Plasmodium spp.
* Severe or complicated malaria including subjects with any of the following:
* Impaired consciousness (eg, obtundation, unarousable coma), seizures or abnormal neurologic exam suggestive of severe or complicated malaria;
* Known hemoglobinuria;
* Jaundice;
* Respiratory distress;
* Persistent vomiting;
* Gross hematuria, as reported by the subject's legally acceptable representative;
* Recent history of convulsions;
* Inability to drink or breastfeed;
* Unable to sit or stand as appropriate for age;
* Known pregnancy or breast-feeding or positive urine pregnancy test (females ≥10 years of age and of child bearing potential);
* History of allergy to or hypersensitivity to azithromycin, any macrolide, chloroquine, artemether, any artemisinin derivative, lumefantrine;
* Any contraindication to any study drug including AZ, CQ and AL;
* History of treatment with any antimalarial drug (such as halofantrine, chloroquine, quinine, mefloquine, Malarone, SP, artemisinin compounds) or antibacterial with known antimalarial activity (macrolides, doxycycline, clindamycin) within 2 weeks prior to enrollment of a subject (and/or of the mother of a subject who is being breastfed) into the study;
* Known or suspected cardiovascular, hepatic or renal abnormality that in the opinion of the investigator would place the subject at increased risk to participate in the study.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 361 (Actual)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Burkina Faso (2):
  - Pfizer Investigational Site, Nouna
  - Pfizer Investigational Site, Ouagadougou
- Pfizer Investigational Site, Abidjan, Côte d’Ivoire
- Pfizer Investigational Site, Navrongo, Ghana
- Pfizer Investigational Site, Kisumu, Kenya
- Mali (2):
  - Pfizer Investigational Site, Bamako, West Africa
  - Pfizer Investigational Site, Sikasso, West Africa

REFERENCES:
- [Derived] Chandra R, Ansah P, Sagara I, Sie A, Tiono AB, Djimde AA, Zhao Q, Robbins J, Penali LK, Ogutu B. Comparison of azithromycin plus chloroquine versus artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria in children in Africa: a randomized, open-label study. Malar J. 2015 Mar 10;14:108. doi: 10.1186/s12936-015-0620-8. PMID 25881046
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661157&StudyName=Azithromycin%20Plus%20Chloroquine%20Versus%20Artemether-Lumefantrine%20For%20The%20Treatment%20Of%20Uncomplicated%20P.%20Falciparum%20Malaria%20In%20Children%20In%20Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 2 age-based Cohorts. Cohort 1=participants between 5-12 years of age, assumed to have some degree of immunity and at less risk for untoward outcome. After demonstration of successful treatment, safety and tolerability in Cohort 1, participants between >=6 months of age to <=59 months of age were enrolled in Cohort 2.
Pre-assignment Details: Participants were enrolled in 2 cohorts based on different age criteria. All participants in Cohort 1 met the age criteria where as 3 participants enrolled in Cohort 2 were slightly older than 5 years (by less than 2 months).
Groups:
- Cohort 1: Azithromycin + Chloroquine: Azithromycin/Chloroquine administered orally once daily for 3 days as a combination tablet (300 milligrams [mg] Azithromycin and 100 mg Chloroquine or 150 mg Azithromycin and 50 mg Chloroquine) on Days 0, 1, 2. The combination tablets were administered on the basis of body weight approximately 30 milligram/kilogram (mg/kg) Azithromycin + approximately 10 mg base/kg Chloroquine base. Cohort 1 included participants between greater than or equal to (>=) 5 years of age and less than or equal to (<=) 12 years of age.
- Cohort 1: Artemether + Lumefantrine: Artemether/Lumefantrine administered orally once daily for 3 days as a combination tablet (20 mg Artemether and 120 mg Lumefantrine) on Days 0, 1, 2. Cohort 1 included participants between >=5 years of age and <=12 years of age.
- Cohort 2: Azithromycin + Chloroquine: Azithromycin/Chloroquine administered orally once daily for 3 days as a combination tablet (300 milligrams [mg] Azithromycin and 100 mg Chloroquine or 150 mg Azithromycin and 50 mg Chloroquine) on Days 0, 1, 2. The combination tablets were administered on the basis of body weight approximately 30 milligram/kilogram (mg/kg) Azithromycin + approximately 10 mg base/kg Chloroquine base. Cohort 2 included participants between >=6 months of age to <=59 months of age.
- Cohort 2: Artemether + Lumefantrine: Artemether/Lumefantrine administered orally once daily for 3 days as a combination tablet (20 mg Artemether and 120 mg Lumefantrine) on Days 0, 1, 2. Cohort 2 included participants between >=6 months of age to <=59 months of age.
Period: Overall Study
Arm/Group | Cohort 1: Azithromycin + Chloroquine | Cohort 1: Artemether + Lumefantrine | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Started | 55 | 51 | 124 | 131
Completed | 51 | 51 | 122 | 128
Not Completed | 4 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 4 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Azithromycin + Chloroquine: Azithromycin/Chloroquine administered orally once daily for 3 days as a combination tablet (300 milligrams [mg] Azithromycin and 100 mg Chloroquine or 150 mg Azithromycin and 50 mg Chloroquine) on Days 0, 1, 2. The combination tablets were administered on the basis of body weight approximately 30 milligram/kilogram (mg/kg) Azithromycin + approximately 10 mg base/kg Chloroquine base. Cohort 1 included participants between >=5 years of age and <=12 years of age.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Azithromycin + Chloroquine | Cohort 1: Artemether + Lumefantrine | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine | Total
Number analyzed (Participants) | 55 | 51 | 124 | 131 | 361
Age, Customized [Number; unit: Participants]
  6 months - less than 5 years | 0 | 0 | 123 | 129 | 252
  5 years - 12 years | 55 | 51 | 1 | 2 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 21 | 50 | 65 | 164
  Male | 27 | 30 | 74 | 66 | 197

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Polymerase Chain Reaction (PCR)-Corrected Adequate Clinical and Parasitologic Response (ACPR) at Day 28 in the Modified Intent-to-treat (mITT) Population
Description: ACPR (PCR-corrected) was defined as asexual Plasmodium falciparum (P.falciparum) parasitologic clearance at Day 28 irrespective of axillary, oral, rectal, or tympanic temperature, without previously meeting the criteria of Early Treatment Failure (ETF) (see measure description in secondary outcome measures 7 and 8) or PCR-corrected Late Treatment Failure (LTF) (which includes PCR-corrected Late Clinical Failures [LCF] - see measure description in secondary outcome measure 9 and 10, and PCR-corrected Late Parasitologic Failures (LPF)- see measure description in secondary outcome measure 11 and 12). PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Day 28
Population: mITT:treated participants who met disease criteria(blood smears positive for P.falciparum monoinfection;asexual parasitemia=1000-100,000 parasites/microliter [mcL];fever/history of fever >=38 degree Celsius[C] [rectal],37.2 degree C [axillary] or >=37.5 degree C [oral] within last 24 hours).Participants in Ivory Coast center excluded from analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 120 | 126
Percentage of participants | 89.27 [82.77 to 95.77] | 98.37 [95.59 to 100.00]
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Null hypothesis: proportion of participants with ACPR (PCR-corrected) of Azithromycin/Chloroquine (AZ-CQ) at Day 28 is less than that of Artemether/Lumefantrine (AL); Alternative hypothesis: proportion of participants with ACPR (PCR-corrected) of AZ-CQ at Day 28 is greater than or equal (non-inferior) to that of AL by a non-inferiority margin of -0.1; Test type: Non-Inferiority or Equivalence — A two-sided 95 percent (%) confidence interval (CI) for the difference in ACPR (PCR corrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR (PCR-corrected) proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. The drug (AZ-CQ) was considered non-inferior with respect to this primary endpoint if the lower bound of this 95% CI was >= -10% points; Kaplan-Meier curves; ACPR percent difference = -9.10, 95% CI 2-sided [-16.02 to -2.18]

2. Primary Outcome: Percentage of Participants With PCR-corrected ACPR at Day 28 in Per-Protocol (PP) Population
Description: ACPR (PCR-corrected) was defined as asexual P.falciparum parasitologic clearance at Day 28 irrespective of axillary, oral, rectal, or tympanic temperature, without previously meeting the criteria of ETF (see measure description in secondary outcome measures 7 and 8) or PCR-corrected LTF (which includes PCR-corrected LCF - see measure description in secondary outcome measure 9 and 10, and PCR-corrected LPF - see measure description in secondary outcome measure 11 and 12). PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Day 28
Population: Per-Protocol (PP) population was a subset of the mITT population, who received all 3 days of study medication to which they were assigned. For ACPR efficacy endpoints, participants in Ivory Coast center excluded from PP population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 114 | 124
Percentage of participants | 93.08 [87.32 to 98.84] | 99.16 [96.97 to 100.00]
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Null hypothesis: proportion of participants with ACPR (PCR-corrected) of AZ-CQ at Day 28 is less than that of AL; Alternative hypothesis: proportion of participants with ACPR (PCR-corrected) of AZ-CQ at Day 28 is greater than or equal (non-inferior) to that of AL by a non-inferiority margin of -0.1; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the difference in ACPR (PCR-corrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR (PCR-corrected) proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. The drug (AZ-CQ) was considered non-inferior with respect to this primary endpoint if the lower bound of this 95% CI was >= -10% points; Kaplan-Meier curves; ACPR percent difference = -6.08, 95% CI 2-sided [-12.10 to -0.05]

3. Secondary Outcome: Percentage of Participants With PCR-corrected ACPR in the mITT Population
Description: ACPR (PCR-corrected) was defined as asexual P.falciparum parasitologic clearance on Days 7, 14, 21, 35, 42 irrespective of axillary, oral, rectal, or tympanic temperature, without previously meeting the criteria of ETF (see measure description in secondary outcome measures 7 and 8) or PCR-corrected LTF (which includes PCR-Corrected LCF- see measure description in secondary outcome measure 9 and 10, and PCR-corrected LPF - see measure description in secondary outcome measure 11 and 12). PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Days 7, 14, 21, 35, 42
Population: mITT population. For ACPR efficacy endpoints, participants in Ivory Coast center excluded from mITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 120 | 126
Percentage of participants
  Day 7 | 94.17 [89.55 to 98.78] | 99.21 [97.25 to 100.00]
  Day 14 | 92.47 [87.30 to 97.64] | 99.21 [97.24 to 100.00]
  Day 21 | 91.59 [86.04 to 97.14] | 98.37 [95.65 to 100.00]
  Day 35 | 89.27 [82.68 to 95.86] | 96.19 [91.85 to 100.00]
  Day 42 | 87.55 [80.08 to 95.03] | 96.19 [91.79 to 100.00]
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-corrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 7; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -5.04, 95% CI 2-sided [-9.93 to -0.15]
Statistical Analysis 2: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-corrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 14; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -6.74, 95% CI 2-sided [-12.15 to -1.32]
Statistical Analysis 3: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-corrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 21; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -6.78, 95% CI 2-sided [-12.82 to -0.75]
Statistical Analysis 4: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-corrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 35; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -6.92, 95% CI 2-sided [-14.59 to 0.76]
Statistical Analysis 5: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-corrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 42; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -8.63, 95% CI 2-sided [-17.08 to -0.18]

4. Secondary Outcome: Percentage of Participants With PCR-corrected ACPR in PP Population
Description: ACPR (PCR-corrected) was defined as asexual P.falciparum parasitologic clearance on Days 7, 14, 21, 35, 42 irrespective of axillary, oral, rectal, or tympanic temperature, without previously meeting the criteria of ETF (see measure description in secondary outcome measures 7 and 8) or PCR-corrected LTF (which includes PCR-corrected LCF - see measure description in secondary outcome measure 9 and 10, and PCR-corrected LPF - see measure description in secondary outcome measure 11 and 12). PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Days 7, 14, 21, 35, 42
Population: PP population. For ACPR efficacy endpoints, participants in Ivory Coast center were excluded from the PP population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 114 | 124
Percentage of participants
  Day 7 | 98.25 [95.39 to 100.00] | 100.00 [NA to NA] — Confidence interval was not calculable as standard error for 100% rate could not be estimated from Kaplan-Meier method.
  Day 14 | 96.46 [92.59 to 100.00] | 100.00 [NA to NA] — Confidence interval was not calculable as standard error for 100% rate could not be estimated from Kaplan-Meier method.
  Day 21 | 95.53 [91.10 to 99.96] | 99.16 [97.03 to 100.00]
  Day 35 | 93.08 [87.22 to 98.95] | 96.96 [92.90 to 100.00]
  Day 42 | 91.29 [84.31 to 98.28] | 96.96 [92.84 to 100.00]
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; Kaplan-Meier, curves; ACPR percent difference = -3.63, 95% CI 2-sided [-8.40 to 1.14]
Statistical Analysis 2: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; Kaplan-Meier, curves; ACPR percent difference = -3.87, 95% CI 2-sided [-10.79 to 3.04]
Statistical Analysis 3: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; Kaplan-Meier, curves; ACPR percent difference = -5.66, 95% CI 2-sided [-13.55 to 2.22]

5. Secondary Outcome: Percentage of Participants With PCR-uncorrected ACPR in the mITT Population
Description: ACPR (PCR-uncorrected) was defined as asexual P.falciparum parasitologic clearance on Days 7, 14, 21, 28, 35, 42 irrespective of axillary, oral, rectal, or tympanic temperature, without previously meeting the criteria of ETF (see measure description in secondary outcome measures 7 and 8) or PCR-uncorrected LTF (which includes PCR-uncorrected LCF - see measure description in secondary outcome measure 9 and 10, and PCR-uncorrected LPF - see measure description in secondary outcome measure 11 and 12). PCR-uncorrected: not adjusted for molecular testing which determined recrudescence or true failures from reinfection.
Time Frame: Days 7, 14, 21, 28, 35, 42
Population: mITT population. For ACPR efficacy endpoints, participants in Ivory Coast center were excluded from mITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 120 | 126
Percentage of participants
  Day 7 | 94.17 [89.55 to 98.78] | 99.21 [97.25 to 100.00]
  Day 14 | 89.08 [83.05 to 95.11] | 96.79 [93.28 to 100.00]
  Day 21 | 67.87 [59.02 to 76.72] | 82.96 [75.91 to 90.01]
  Day 28 | 51.55 [42.07 to 61.02] | 73.31 [65.10 to 81.52]
  Day 35 | 44.67 [35.24 to 54.11] | 62.91 [54.00 to 71.82]
  Day 42 | 37.80 [28.58 to 47.02] | 56.29 [47.12 to 65.46]
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-uncorrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 7; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -5.04, 95% CI 2-sided [-9.93 to -0.15]
Statistical Analysis 2: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-uncorrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 14; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -7.71, 95% CI 2-sided [-14.54 to -0.88]
Statistical Analysis 3: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-uncorrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 21; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -15.09, 95% CI 2-sided [-26.24 to -3.94]
Statistical Analysis 4: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-uncorrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 28; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -21.76, 95% CI 2-sided [-34.14 to -9.39]
Statistical Analysis 5: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-uncorrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 35; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -18.24, 95% CI 2-sided [-31.05 to -5.43]
Statistical Analysis 6: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-uncorrected) proportions [(AZ-CQ)-(AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the greenwood formula. Estimates for Day 42; Test type: Superiority or Other; Kaplan-Meier curves; ACPR Percent difference = -18.49, 95% CI 2-sided [-31.33 to -5.65]

6. Secondary Outcome: Percentage of Participants With PCR-uncorrected ACPR in PP Population
Description: as for outcome 5
Time Frame: Days 7, 14, 21, 28, 35, 42
Population: PP population. For ACPR efficacy endpoints, participants in Ivory Coast center were excluded from the PP population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 114 | 124
Percentage of participants
  Day 7 | 98.25 [95.39 to 100.00] | 100.00 [NA to NA] — Confidence interval not calculable when rate is 100%.
  Day 14 | 92.89 [87.69 to 98.08] | 97.56 [94.42 to 100.00]
  Day 21 | 70.56 [61.67 to 79.45] | 83.62 [76.65 to 90.60]
  Day 28 | 54.28 [44.57 to 63.98] | 73.90 [65.71 to 82.08]
  Day 35 | 47.04 [37.31 to 56.77] | 63.41 [54.49 to 72.34]
  Day 42 | 39.80 [30.24 to 49.36] | 56.74 [47.54 to 65.94]
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -4.67, 95% CI 2-sided [-10.60 to 1.25]
Statistical Analysis 2: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -13.07, 95% CI 2-sided [-24.21 to -1.92]
Statistical Analysis 3: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -19.62, 95% CI 2-sided [-32.16 to -7.08]
Statistical Analysis 4: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; Kaplan-Meier curves; ACPR percent difference = -16.38, 95% CI 2-sided [-29.42 to -3.33]
Statistical Analysis 5: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; A two-sided 95% CI for the difference in ACPR (PCR-uncorrected) proportions [(AZ-CQ)- (AL)] using the normal approximation to the binomial with continuity correction was constructed based on the estimated ACPR proportions from the Kaplan-Meier curves and their standard errors estimated by the Greenwood formula. Estimates for Day 42; Test type: Superiority or Other; Kaplan-Meier curves; ACPR Percent difference = -16.94, 95% CI 2-sided [-30.04 to -3.83]

7. Secondary Outcome: Percentage of Participants With Early Treatment Failure (ETF) in the mITT Population (PCR-corrected)
Description: ETF defined as participants who met the following criteria:
  1. Developed signs of severe malaria or clinical deterioration that required rescue medication on Days 0, 1, 2 or 3, in the presence of P. falciparum parasitemia
  2. Last available asexual P. falciparum parasite count on Day 2 greater than the first available parasite count on Day 0 (Baseline), irrespective of axillary, oral or rectal temperature.
  3. Parasitemia (P. falciparum) on Day 3 with fever or
  4. Last available P. falciparum parasite count on Day 3 >=25% of the first available parasite count on Day 0 (Baseline).
  PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Day 0 up to Day 3
Population: mITT population, participants in Ivory Coast center were excluded from mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 120 | 126
Percentage of participants | 5.83 | 0.79

8. Secondary Outcome: Percentage of Participants With ETF in PP Population (PCR-corrected)
Description: ETF defined as participants who met the following criteria:
  1. Developed signs of severe malaria or clinical deterioration that required rescue medication on Days 0, 1, 2 or 3, in the presence of P.falciparum parasitemia
  2. Last available asexual P.falciparum parasite count on Day 2 greater than the first available parasite count on Day 0 (Baseline), irrespective of axillary, oral or rectal temperature.
  3. Parasitemia (P.falciparum) on Day 3 with fever or
  4. Last available P.falciparum parasite count on Day 3 >=25% of the first available parasite count on Day 0 (Baseline).
  PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Day 0 up to Day 3
Population: PP population, participants in Ivory Coast center were excluded from the PP population.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 114 | 124
Percentage of participants | 1.75 | 0

9. Secondary Outcome: Percentage of Participants With Late Clinical Failure (LCF) in the mITT Population (PCR-corrected)
Description: LCF included participants who met any of the following criteria:
  1. Development of signs of severe malaria or clinical deterioration requiring rescue medication after Day 3 in the presence of P.falciparum parasitemia, without previously meeting any of the criteria of ETF (see measure description in secondary outcome measures 7 and 8)
  2. Presence of P.falciparum parasitemia and fever on any day from Day 4 onward, without previously meeting any of the criteria of ETF (see measure description in secondary outcome measures 7 and 8). PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Days 7, 14, 21, 28, 35, 42
Population: mITT population, participants in Ivory Coast center were excluded from mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 120 | 126
Percentage of participants
  Day 7 | 0 | 0
  Day 14 | 0 | 0
  Day 21 | 0 | 0
  Day 28 | 0 | 0
  Day 35 | 0 | 0
  Day 42 | 0 | 0

10. Secondary Outcome: Percentage of Participants With LCF in PP Population (PCR-corrected)
Description: as for outcome 9
Time Frame: Days 7, 14, 21, 28, 35, 42
Population: PP population, participants in Ivory Coast center were excluded from the PP population.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 114 | 124
Percentage of participants
  Day 7 | 0 | 0
  Day 14 | 0 | 0
  Day 21 | 0 | 0
  Day 28 | 0 | 0
  Day 35 | 0 | 0
  Day 42 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Late Parasitologic Failure (LPF) in the mITT Population (PCR-corrected)
Description: LPF: Presence of P. falciparum parasitemia in the mITT population on any day from Day 7 onward and the absence of fever without previously meeting any of the criteria of ETF (see measure description in secondary outcome measures 7 and 8) or LCF (see measure description in secondary outcome measure 9 and 10). PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Days 7, 14, 21, 28, 35, 42
Population: mITT population, participants in Ivory Coast center were excluded from mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 120 | 126
Percentage of participants
  Day 7 | 0 | 0
  Day 14 | 1.67 | 0
  Day 21 | 2.50 | 0.79
  Day 28 | 4.17 | 0.79
  Day 35 | 4.17 | 2.38
  Day 42 | 5.00 | 2.38

12. Secondary Outcome: Percentage of Participants With LPF in PP Population (PCR-corrected)
Description: LPF: Presence of P.falciparum parasitemia in the PP population on any day from Day 7 onward and the absence of fever without previously meeting any of the criteria of ETF (see measure description in secondary outcome measures 7 and 8) or LCF (see measure description in secondary outcome measure 9 and 10). PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Days 7, 14, 21, 28, 35, 42
Population: PP population, participants in Ivory Coast center were excluded from the PP population.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 114 | 124
Percentage of participants
  Day 7 | 0 | 0
  Day 14 | 1.75 | 0
  Day 21 | 2.63 | 0.81
  Day 28 | 4.39 | 0.81
  Day 35 | 4.39 | 2.42
  Day 42 | 5.26 | 2.42

13. Secondary Outcome: Percentage of Participants With Asexual Parasitologic Response (PCR-corrected)
Description: Percentage of participants who were cleared of asexual parasites. Asexual parasite clearance - clearance of asexual P.falciparum parasitemia within 7 days of initiation of treatment without subsequent recurrence (PCR-corrected) through the day of consideration. PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Day 7, 14, 21, 28, 35, 42
Population: mITT population. Number of participants analyzed (N)=participants with evaluable data, including participants in the Ivory Coast center. "n"=participants who were evaluable at specified time points for each arm, respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 120 | 128
Percentage of participants
  Day 7 (n=120, 128) | 93.33 | 99.22
  Day 14 (n=120, 127) | 91.67 | 99.21
  Day 21 (n=120, 128) | 90.83 | 98.44
  Day 28 (n=120, 127) | 89.17 | 98.43
  Day 35 (n=120, 128) | 89.17 | 96.88
  Day 42 (n=120, 127) | 88.33 | 96.85
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 7; Test type: Superiority or Other; large sample approximation to binomial; percent difference = -5.89, 95% CI 2-sided [-11.02 to -0.75]
Statistical Analysis 2: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 14; Test type: Superiority or Other; large sample approximation to binomial; percent difference = -7.55, 95% CI 2-sided [-13.14 to -1.95]
Statistical Analysis 3: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 21; Test type: Superiority or Other; large sample approximation to binomial; percent difference = -7.60, 95% CI 2-sided [-13.61 to -1.60]
Statistical Analysis 4: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 28; Test type: Superiority or Other; Large sample approximation to binomial; percent difference = -9.26, 95% CI 2-sided [-15.64 to -2.87]
Statistical Analysis 5: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 35; Test type: Superiority or Other; Large sample approximation to binomial; percent difference = -7.71, 95% CI 2-sided [-14.45 to -0.97]
Statistical Analysis 6: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 42; Test type: Superiority or Other; Large sample approximation to binomial; percent difference = -8.52, 95% CI 2-sided [-15.43 to -1.60]

14. Secondary Outcome: Percentage of Participants With Gametocytologic Response
Description: Gametocyte response/absence/clearance: Clearance of P.falciparum gametocytemia (PCR-uncorrected) (attainment of 2 consecutive zero gametocyte counts) without subsequent recurrence through the day of consideration. PCR-uncorrected: not adjusted for molecular testing which determined recrudescence or true failures from reinfection.
Time Frame: Days 7, 14, 21, 28, 35, 42
Population: mITT population. "N"= participants with evaluable data, including participants in the Ivory Coast center. "n"=participants who were evaluable at specified time points for each arm, respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 122 | 130
Percentage of participants
  Day 7 (n=122, 129) | 81.97 | 91.47
  Day 14 (n=122, 130) | 81.15 | 91.54
  Day 21 (n=122, 130) | 80.33 | 93.08
  Day 28 (n=122, 130) | 81.97 | 93.08
  Day 35 (n=122, 130) | 81.97 | 92.31
  Day 42 (n=122, 130) | 80.33 | 91.54
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 7; Test type: Superiority or Other; Large sample approximation to binomial; percent difference = -9.51, 95% CI 2-sided [-18.27 to -0.74]
Statistical Analysis 2: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 14; Test type: Superiority or Other; Large sample approximation to binomial; percent difference = -10.39, 95% CI 2-sided [-19.23 to -1.55]
Statistical Analysis 3: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 21; Test type: Superiority or Other; Large sample approximation to binomial; percent difference = -12.75, 95% CI 2-sided [-21.45 to -4.04]
Statistical Analysis 4: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 28; Test type: Superiority or Other; Large sample approximation to binomial; percent difference = -11.11, 95% CI 2-sided [-19.62 to -2.60]
Statistical Analysis 5: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 35; Test type: Superiority or Other; Large sample approximation to binomial; percent difference = -10.34, 95% CI 2-sided [-18.97 to -1.71]
Statistical Analysis 6: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Day 42; Test type: Superiority or Other; Large sample approximation to binomial; percent difference = -11.21, 95% CI 2-sided [-20.14 to -2.28]

15. Secondary Outcome: Fever Clearance Time
Description: Calculated as time of first occurrence of two consecutive time points with temperature less than (<) 38.0 degrees C/100.4 degrees Fahrenheit (F) (rectal), 37.2 degrees C/99.0 degrees F (axillary), or <37.5 degrees C/99.5 degrees F (oral).
Time Frame: Baseline to Day 42
Population: mITT population, including participants in the Ivory Coast center.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 124 | 131
Hours | 24.000 [1 to 504] | 24.000 [1 to 336]
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Time to event data was analyzed using the Kaplan-Meier curve; Test type: Superiority or Other; p = 0.2564, Kaplan-Meier, log rank

16. Secondary Outcome: Asexual Plasmodium Falciparum Parasite Clearance Time
Description: Defined as time to first of two consecutive zero asexual P. falciparum parasite (PCR-corrected) counts, regardless of recurrence of parasitemia later. PCR-corrected refers to the use of molecular testing to differentiate recrudescence from reinfection in the context of an efficacy evaluation.
Time Frame: Baseline to Day 42
Population: mITT population, including participants in the Ivory Coast center.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 124 | 131
Hours | 48.000 [24 to 504] | 24.000 [1 to 48]
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Time to event data was analyzed using the Kaplan-Meier curve; Test type: Superiority or Other; p < 0.0001, Kaplan-Meier, log rank

17. Secondary Outcome: Nadir Hemoglobin Level
Description: Nadir hemoglobin for each participant was defined as the minimum hemoglobin values obtained from Day 0 through Day 3.
Time Frame: Day 0 through Day 3
Population: mITT population, including participants in the Ivory Coast center.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 124 | 131
grams per deciliter (g/dL) | 9.63 (1.53) | 9.82 (1.61)

18. Secondary Outcome: Change From Nadir Hemoglobin Level at Days 14, 28, and 42
Description: Change from nadir = observation minus nadir. Nadir defined as the minimum value for each participant on Days 0-3.
Time Frame: Day 14, 28, 42
Population: mITT population. "N" = number of participants with evaluable data, including participants in the Ivory Coast center. "n"=participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 122 | 128
g/dL
  Change at Day 14 (n=122, 127) | 0.52 (0.11) | 0.44 (0.13)
  Change at Day 28 (n=122, 127) | 1.15 (0.11) | 0.96 (0.13)
  Change at Day 42 (n=122, 128) | 1.29 (0.12) | 1.14 (0.14)

19. Secondary Outcome: Time to Recurrence of Parasitemia
Description: Time from the day of clearance to the time of recurrence of asexual P.falciparum parasitemia (PCR-uncorrected).
Time Frame: Baseline (Day 0) to Day 42
Population: mITT population, including participants in the Ivory Coast center.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 124 | 131
Days | 34 [2 to 42] | NA [7 to 43] — Median time to recurrence could not be calculated for participants in the Artemether-Lumefantrine treatment groups since fewer than 50% of the participants experienced recurrent parasitemia during the study.
Statistical Analysis 1: Comparison: Cohort 2: Azithromycin + Chloroquine vs Cohort 2: Artemether + Lumefantrine; Time to event data was analyzed using the Kaplan-Meier curve; Test type: Superiority or Other; p = 0.0006, Kaplan-Meier, log rank

20. Secondary Outcome: Number of Participants With Recurrent Parasitemia Versus Baseline Plasmodium Falciparum Chloroquine Resistance Transporter (PfCRT) Status
Time Frame: Baseline to Day 42
Population: Data for this outcome measure was not analyzed as per change in planned analysis.
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Percentage of Participants With PfCRT in True Failures
Description: A genetic marker, P.falciparum chloroquine resistance transporter (PfCRT), indicative of P.falciparum chloroquine resistance was to be determined from blood blots obtained on Day 0 and at the time of treatment failure. Treatment failure was defined as any of the following events that a participant experienced from Day 0 through the Day 42 visit: ETF (see measure description in secondary outcome measures 7 and 8), LCF (PCR corrected) (see measure description in secondary outcome measure 9 and 10), or LPF (PCR corrected) (see measure description in secondary outcome measure 11 and 12). Recrudescence of asexual P.falciparum parasites was considered treatment failure.
Time Frame: Baseline to Day 42
Population: Data for this outcome measure was not analyzed as per change in planned analysis.
Arm/Group | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Cohort 1: Azithromycin + Chloroquine: Azithromycin/Chloroquine administered orally once daily for 3 days as a combination tablet (300 milligrams [mg] Azithromycin and 100 mg Chloroquine or 150 mg Azithromycin and 50 mg Chloroquine) on Days 0, 1, 2. The combination tablets were administered on the basis of body weight approximately 30 milligram/kilogram (mg/kg) Azithromycin + approximately 10 mg base/kg Chloroquine base). Cohort 1 included participants between >=5 years of age and <=12 years of age.
Arm/Group | Cohort 1: Azithromycin + Chloroquine | Cohort 1: Artemether + Lumefantrine | Cohort 2: Azithromycin + Chloroquine | Cohort 2: Artemether + Lumefantrine
Serious Adverse Events (participants affected / at risk) | 1/55 | 2/51 | 0/124 | 1/131
Other Adverse Events (participants affected / at risk) | 40/55 | 36/51 | 103/124 | 99/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Azithromycin + Chloroquine (N=55) | Cohort 1: Artemether + Lumefantrine (N=51) | Cohort 2: Azithromycin + Chloroquine (N=124) | Cohort 2: Artemether + Lumefantrine (N=131)
Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 0
Malaria (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Azithromycin + Chloroquine (N=55) | Cohort 1: Artemether + Lumefantrine (N=51) | Cohort 2: Azithromycin + Chloroquine (N=124) | Cohort 2: Artemether + Lumefantrine (N=131)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 3 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 0 | 0
Conjunctival pallor (Eye disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 3 | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 5 | 4 | 14
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4 | 8
Nausea (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 11 | 5 | 38 | 13
Chills (General disorders) | 2 | 2 | 3 | 5
Fatigue (General disorders) | 1 | 2 | 0 | 3
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 3 | 2
Pyrexia (General disorders) | 4 | 3 | 17 | 27
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 1
Body tinea (Infections and infestations) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 4 | 9
Dysentery (Infections and infestations) | 0 | 1 | 1 | 1
Giardiasis (Infections and infestations) | 0 | 1 | 0 | 0
Infection parasitic (Infections and infestations) | 14 | 11 | 37 | 31
Malaria (Infections and infestations) | 5 | 4 | 26 | 19
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 1 | 2 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Tinea capitis (Infections and infestations) | 5 | 2 | 2 | 2
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 9 | 12
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 9 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 | 5 | 4 | 4
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 15 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 1 | 8 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 3
Inflammation (General disorders) | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 1
Product taste abnormal (General disorders) | 0 | 0 | 1 | 0
Amoebiasis (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 1
Blister infected (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 2
Furuncle (Infections and infestations) | 0 | 0 | 1 | 5
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 5
Helminthic infection (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1
Mumps (Infections and infestations) | 0 | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 8
Septic rash (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Viral rash (Infections and infestations) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Cohort 1 was a screening cohort, meant for safety evaluation, but not included in the efficacy assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.